CLINICAL TRIAL: NCT07353047
Title: The Efficacy of Personalized Local Anesthetic Dosing Based on Ultrasound-Measured Nerve Cross-Sectional Area in Brachial Plexus Block: a Non-Inferiority Randomized Controlled Trial.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Ju Gao, Study Director, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2025ky401
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Upper Limb Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CSA-based Dosing Group (Experimental): The cross-sectional area (CSA) of the brachial plexus nerves at the interscalene groove is measured using ultrasound in the short-axis view.
  The dose of 0.5% ropivacaine is calculated individually using the formula: Volume (mL) = CSA (mm²) × Conversion Coefficient (mL/mm²). The conversion coefficient is derived from a pilot dose-finding study conducted prior to the main trial.
  The total dose for any participant will not exceed the maximum recommended safe dose of ropivacaine (≤225 mg).
  The nerve block is performed under ultrasound guidance by an experienced anesthesiologist.
  Interventions: Drug: CSA-based dosing of Ropivacaine
- Experience-based Dosing Group (Other): The dose of 0.5% ropivacaine is determined solely by the clinical judgment and experience of the attending anesthesiologist, reflecting common real-world practice.The nerve block is performed under ultrasound guidance by an experienced anesthesiologist.
  Interventions: Drug: Experience-based dosing of Ropivacaine
- Weight-based Dosing Group (Other): The dose of 0.5% ropivacaine is calculated based on the participant's body weight using a standard formula: Dose (mg) = 2.5 mg/kg.
  The corresponding volume is then administered. The nerve block is performed under ultrasound guidance by an experienced anesthesiologist.
  Interventions: Drug: Weight-based dosing of Ropivacaine

INTERVENTIONS:
Drug: CSA-based dosing of Ropivacaine — Participants assigned to this group will receive an ultrasound-guided interscalene brachial plexus block. First, the cross-sectional area (CSA) of the brachial plexus nerves at the interscalene groove will be measured in the short-axis view using ultrasound. The dose of 0.5% ropivacaine will then be calculated individually using the formula: Volume (mL) = CSA (mm²) × K, where K is a conversion coefficient (in mL/mm²) determined from a prior pilot dose-finding study. The total administered dose will not exceed the maximum recommended safe dose of ropivacaine (225 mg). The block will be performed by an experienced anesthesiologist under real-time ultrasound guidance.
  Arms: CSA-based Dosing Group
Drug: Experience-based dosing of Ropivacaine — Participants assigned to this group will receive an ultrasound-guided interscalene brachial plexus block. The volume of 0.5% ropivacaine to be injected will be determined solely by the clinical judgment and experience of the attending anesthesiologist, reflecting standard real-world practice. The total administered dose will not exceed the maximum recommended safe dose of ropivacaine (225 mg). The block will be performed by an experienced anesthesiologist under real-time ultrasound guidance.
  Arms: Experience-based Dosing Group
Drug: Weight-based dosing of Ropivacaine — Participants assigned to this group will receive an ultrasound-guided interscalene brachial plexus block. The dose of 0.5% ropivacaine will be calculated based on the participant's body weight using the standard formula: Dose (mg) = 2.5 mg/kg. The corresponding volume will then be administered. The total administered dose will not exceed the maximum recommended safe dose of ropivacaine (225 mg). The block will be performed by an experienced anesthesiologist under real-time ultrasound guidance.
  Arms: Weight-based Dosing Group

SUMMARY:
This is a prospective, randomized, assessor-blinded, three-arm, non-inferiority clinical trial. The study aims to compare the effectiveness and safety of an individualized dosing strategy for local anesthetic in brachial plexus blocks against two standard methods. The experimental intervention uses ultrasound to measure the cross-sectional area (CSA) of the brachial plexus nerves to calculate a patient-specific dose of 0.5% ropivacaine. This is compared to a standard weight-based dosing regimen (2.5 mg/kg) and dosing based on the anesthesiologist's clinical experience. A total of 350 adult patients scheduled for elective unilateral upper limb surgery will be randomly assigned to one of the three groups. The primary outcome is the success rate of the nerve block 30 minutes after administration. Secondary outcomes include assessments of diaphragmatic function, postoperative pain scores, the incidence of complications (such as nerve involvement or systemic toxicity), and patient satisfaction. The hypothesis is that the CSA-based dosing method will be non-inferior to the conventional methods in achieving successful anesthesia while potentially optimizing drug dosage.

ELIGIBILITY:
Inclusion Criteria:

Age 18-80 years old, proposed for elective unilateral upper extremity surgery; ASA grade I-III; Planned to undergo ultrasound-guided interscalene sulcus brachial plexus block; Normal preoperative respiratory function; No history of neck surgery; No use of drugs that affect nerve conduction or opioids within 30 days prior to surgery

Exclusion Criteria:

Local infection, coagulation dysfunction, neuropathy; Allergy to ropivacaine or amide local anesthetics; Severe hepatic and renal insufficiency; Pregnancy or lactation; Expected dosing required to exceed the maximum safe single safe dose of ropivacaine; Inability to cooperate with ultrasound measurements or nerve block operators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Block Success Rate | At 30 minutes after block completion

CONTACTS AND LOCATIONS:
Locations (1):
- Jianjun Qian, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No